CLINICAL TRIAL: NCT00708760
Title: Moderate Sedation Education Software
Brief Title: Moderate Sedation Educational Software
Status: Terminated | Type: Observational
Why Stopped: Vastly under enrolled due to delays in software development
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 23011; University of Utah VIP grant
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2012-03

CONDITIONS: Moderate Sedation Training
Keywords: web based learning; moderate sedation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2: web based learning group
  Interventions: Behavioral: web based training
- 1: paper based learning group
  Interventions: Behavioral: paper based training

INTERVENTIONS:
Behavioral: paper based training — read selected material, test skills learned in simulator lab
  Groups: 1
Behavioral: web based training — read and view selected web based material, test skills learned in simulator lab
  Groups: 2

SUMMARY:
We propose to develop and evaluate an interactive education software for administering moderate sedation by non-anesthesiologists.

DETAILED DESCRIPTION:
The course will be founded upon JCAHO's and ASA's guidelines for sedation, emphasizing the concepts with animations, audio, scenarios, and quizzes. Interactive feedback will be incorporated to guide the clinician during the course. The course will be offered commercially over the World Wide Web, with successful completion providing continuing medical education (CME) credit. It will fulfill JCAHO recommended guidelines. In a controlled simulated environment, the hypothesis that the web based training protocol will provide the practitioner the knowledge base necessary to manage the four scenarios as well or better than practitioners completing the standard moderate sedation certification course will be tested.

1) Evaluate the effectiveness of the course. The University of Utah Center for Patient Simulation is an ideal environment to evaluate the efficacy of a web-based training course. The new web-based course will be compared to standard course material and lessons. We will recruit 40 nurses who administer moderate sedation at the University of Utah Health Sciences Center. Half of the nurses will receive traditional training (typical course and guidelines published from the literature), and half will receive the web-based course. Users will be tested on their knowledge of moderate sedation with four moderate sedation scenarios, in which the simulated patient experiences over-sedation, apnea, and excessive pain.

ELIGIBILITY:
Inclusion Criteria:

* general nursing staff at the University of Utah
* currently required to obtain moderate sedation training
* an equal basis all clinicians in the respective departments

Exclusion Criteria:

* nurses and other personnel who do not administer moderate sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: nurses providing moderate sedation
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-04; Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

PRIMARY OUTCOMES:
to determine which group - web based or paper based is more effective | at the end of simulation

CONTACTS AND LOCATIONS:
Overall Officials: James Agutter, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States